CLINICAL TRIAL: NCT06367049
Title: Methylation-specific PCR Test for Early Screening and Early Diagnosis of Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Women and Children Hospital (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, YiJun Hua, Chief Physician, Sun Yat-sen University
Other Study IDs: 2023-FXY-230-NPC
Record Dates: First submitted 2024-03-27; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma; Early Diagnosis of Cancer
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retained biospecimens include nasopharyngeal swab specimens and peripheral blood specimens.

GROUPS / COHORTS (2):
- Patient group: Sampling their nasopharyngeal swab specimens and peripheral blood specimens.
  Interventions: Diagnostic Test: Methylation-specific PCR
- Non-patient group: Sampling their nasopharyngeal swab specimens and peripheral blood specimens.
  Interventions: Diagnostic Test: Methylation-specific PCR

INTERVENTIONS:
Diagnostic Test: Methylation-specific PCR — Methylation-specific PCR is the simplest and quickest method for qualitative detection of methylation status.
  The unmethylated C base is converted to U by bisulfite conversion, which is subsequently amplified by PCR with primers (methylation-specific and non-methylation-specific primers) and subsequently detected by agarose gel electrophoresis or a probe. The key to MSP is to design PCR primers for specific gene regions. The research team of this project has previously found the sequence sites of methylation of H4C6, Septin9 and RASSF1A genes in nasopharyngeal carcinoma tissues through methylation sequencing, and designed specific MSP amplification primers and probes accordingly, which can perform methylation detection easily and quickly.

SUMMARY:
Nasopharyngeal carcinoma is one of the most common malignant tumors in China, with the progress of radiochemical comprehensive treatment, early stage The 5-year survival rate of nasopharyngeal cancer is more than 95%. However, due to the hidden site of nasopharyngeal carcinoma and the lack of obvious early clinical symptoms, more than 70% of the 87,000 newly diagnosed cases each year belong to the advanced stage of nasopharyngeal carcinoma, and the 5-year survival rate of advanced nasopharyngeal carcinoma is only about 70%. Therefore, early screening and diagnosis and early treatment are the key to improve the survival of patients with nasopharyngeal cancer. Selecting a sensitive and accurate biomarker for nasopharyngeal cancer and relying on a simple and feasible examination method for sampling detection will greatly improve the early diagnosis rate of nasopharyngeal cancer.

DNA methylation is a form of chemical modification of DNA that can be done without altering the DNA sequence changes in genetic expression. The main role of DNA methylation is to regulate gene expression. Tumor suppressor genes play the functions of regulating cell differentiation, maturation and programmed death. However, if methylation of promoter region occurs, the expression of tumor suppressor genes is inhibited and the function is lost, resulting in cells remaining in the stage of low differentiation and proliferation, inhibition of apoptosis, formation of blood vessels by cluster cells, loss of cell adhesion, and formation of tumors. It can be seen that DNA methylation occurs in the early stage of tumor, and this biological feature makes it a strong application prospect in early tumor screening.

There are many methods to detect DNA Methylation, among which methylation-specific PCR (MSP) can easily and quickly determine the methylation status of a specific gene, meeting the affordable, convenient, and easy to generalize characteristics required for screening tests. In combination with previous MSP experiments and previous reports, we found that the methylation levels of promoter fragments of H4C6, Septin9 and RASSF1A genes in nasopharyngeal carcinoma tissues were significantly higher than those in healthy human nasopharyngeal tissues. This suggests that methylation of these three genes may be used as biomarkers for early screening and diagnosis of nasopharyngeal carcinoma.

Therefore, this study intends to detect the methylation status of H4C6, Septin9 and RASSF1A genes based on MSP method with simple operation and low cost. Using clinicopathological diagnosis as the gold standard, the value of this gene methylation index in early screening and early diagnosis of nasopharyngeal cancer was verified, providing a new detection index and method for improving the early diagnosis rate of nasopharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Case group (nasopharyngeal carcinoma group): nasopharyngeal carcinoma confirmed by histology or cytology. Control group (non-nasopharyngeal carcinoma group): no nasopharyngeal carcinoma subjects.
2. Age ≥18 years and ≤70 years.
3. No previous history of other tumors, and no current tumors.

Exclusion Criteria:

1. Karnofsky score ≤70 points or Zubrod score >2 points.
2. There are serious medical complications, dysfunction of important organs (heart, lung, liver, kidney) or neuropsychiatric disorders.
3. Other patients or volunteers deemed unsuitable for inclusion by the supervising physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects in the case group (nasopharyngeal carcinoma group) and the control group (non-nasopharyngeal carcinoma group) are from Sun Yat-sen University Cancer Hosptial, Guangdong Women and Children Hospital and Tumor Hospital of Guangzhou Medical College.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | through study completion, an average of 1 year
  The proportion of patients with pathological diagnosis of nasopharyngeal carcinoma with positive methylation index.

SECONDARY OUTCOMES:
Specificity | through study completion, an average of 1 year
  The proportion of non-nasopharyngeal carcinoma patients with negative methylation index.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jun Hua, Phd, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karimi M, Johansson S, Stach D, Corcoran M, Grander D, Schalling M, Bakalkin G, Lyko F, Larsson C, Ekstrom TJ. LUMA (LUminometric Methylation Assay)--a high throughput method to the analysis of genomic DNA methylation. Exp Cell Res. 2006 Jul 1;312(11):1989-95. doi: 10.1016/j.yexcr.2006.03.006. Epub 2006 Apr 19. PMID 16624287
- [Background] Lyu JY, Chen JY, Zhang XJ, Zhang MW, Yu GS, Zhang L, Wen Z. Septin 9 Methylation in Nasopharyngeal Swabs: A Potential Minimally Invasive Biomarker for the Early Detection of Nasopharyngeal Carcinoma. Dis Markers. 2020 May 5;2020:7253531. doi: 10.1155/2020/7253531. eCollection 2020. PMID 32454907
- [Background] Chang HW, Chan A, Kwong DL, Wei WI, Sham JS, Yuen AP. Evaluation of hypermethylated tumor suppressor genes as tumor markers in mouth and throat rinsing fluid, nasopharyngeal swab and peripheral blood of nasopharygeal carcinoma patient. Int J Cancer. 2003 Jul 20;105(6):851-5. doi: 10.1002/ijc.11162. PMID 12767073
- [Background] Wong TS, Kwong DL, Sham JS, Wei WI, Kwong YL, Yuen AP. Quantitative plasma hypermethylated DNA markers of undifferentiated nasopharyngeal carcinoma. Clin Cancer Res. 2004 Apr 1;10(7):2401-6. doi: 10.1158/1078-0432.ccr-03-0139. PMID 15073117
- [Background] Hutajulu SH, Indrasari SR, Indrawati LP, Harijadi A, Duin S, Haryana SM, Steenbergen RD, Greijer AE, Middeldorp JM. Epigenetic markers for early detection of nasopharyngeal carcinoma in a high risk population. Mol Cancer. 2011 May 2;10:48. doi: 10.1186/1476-4598-10-48. PMID 21535891
- [Background] Ye M, Huang T, Ni C, Yang P, Chen S. Diagnostic Capacity of RASSF1A Promoter Methylation as a Biomarker in Tissue, Brushing, and Blood Samples of Nasopharyngeal Carcinoma. EBioMedicine. 2017 Apr;18:32-40. doi: 10.1016/j.ebiom.2017.03.038. Epub 2017 Apr 2. PMID 28396012
- [Background] Li Y, Yang X, Du X, Lei Y, He Q, Hong X, Tang X, Wen X, Zhang P, Sun Y, Zhang J, Wang Y, Ma J, Liu N. RAB37 Hypermethylation Regulates Metastasis and Resistance to Docetaxel-Based Induction Chemotherapy in Nasopharyngeal Carcinoma. Clin Cancer Res. 2018 Dec 15;24(24):6495-6508. doi: 10.1158/1078-0432.CCR-18-0532. Epub 2018 Aug 21. PMID 30131385
- [Background] Shi F, Zhou M, Shang L, Du Q, Li Y, Xie L, Liu X, Tang M, Luo X, Fan J, Zhou J, Gao Q, Qiu S, Wu W, Zhang X, Bode AM, Cao Y. EBV(LMP1)-induced metabolic reprogramming inhibits necroptosis through the hypermethylation of the RIP3 promoter. Theranostics. 2019 Apr 13;9(9):2424-2438. doi: 10.7150/thno.30941. eCollection 2019. PMID 31131045
- [Background] Zhao Y, Hong XH, Li K, Li YQ, Li YQ, He SW, Zhang PP, Li JY, Li Q, Liang YL, Chen Y, Ma J, Liu N, Chen YP. ZNF582 hypermethylation promotes metastasis of nasopharyngeal carcinoma by regulating the transcription of adhesion molecules Nectin-3 and NRXN3. Cancer Commun (Lond). 2020 Dec;40(12):721-737. doi: 10.1002/cac2.12104. Epub 2020 Oct 10. PMID 33038291
- [Background] Chen Y, Zhao Y, Yang X, Ren X, Huang S, Gong S, Tan X, Li J, He S, Li Y, Hong X, Li Q, Ding C, Fang X, Ma J, Liu N. USP44 regulates irradiation-induced DNA double-strand break repair and suppresses tumorigenesis in nasopharyngeal carcinoma. Nat Commun. 2022 Jan 25;13(1):501. doi: 10.1038/s41467-022-28158-2. PMID 35079021
- [Background] Papanicolau-Sengos A, Aldape K. DNA Methylation Profiling: An Emerging Paradigm for Cancer Diagnosis. Annu Rev Pathol. 2022 Jan 24;17:295-321. doi: 10.1146/annurev-pathol-042220-022304. Epub 2021 Nov 4. PMID 34736341
- [Background] Roy D, Tiirikainen M. Diagnostic Power of DNA Methylation Classifiers for Early Detection of Cancer. Trends Cancer. 2020 Feb;6(2):78-81. doi: 10.1016/j.trecan.2019.12.006. Epub 2020 Feb 3. PMID 32061307
- [Background] Widschwendter M, Zikan M, Wahl B, Lempiainen H, Paprotka T, Evans I, Jones A, Ghazali S, Reisel D, Eichner J, Rujan T, Yang Z, Teschendorff AE, Ryan A, Cibula D, Menon U, Wittenberger T. The potential of circulating tumor DNA methylation analysis for the early detection and management of ovarian cancer. Genome Med. 2017 Dec 22;9(1):116. doi: 10.1186/s13073-017-0500-7. PMID 29268796
- [Background] Sung CK, Yim H. CRISPR-mediated promoter de/methylation technologies for gene regulation. Arch Pharm Res. 2020 Jul;43(7):705-713. doi: 10.1007/s12272-020-01257-8. Epub 2020 Jul 28. PMID 32725389
- [Background] Mattei AL, Bailly N, Meissner A. DNA methylation: a historical perspective. Trends Genet. 2022 Jul;38(7):676-707. doi: 10.1016/j.tig.2022.03.010. Epub 2022 Apr 30. PMID 35504755
- [Background] Ji MF, Sheng W, Cheng WM, Ng MH, Wu BH, Yu X, Wei KR, Li FG, Lian SF, Wang PP, Quan W, Deng L, Li XH, Liu XD, Xie YL, Huang SJ, Ge SX, Huang SL, Liang XJ, He SM, Huang HW, Xia SL, Ng PS, Chen HL, Xie SH, Liu Q, Hong MH, Ma J, Yuan Y, Xia NS, Zhang J, Cao SM. Incidence and mortality of nasopharyngeal carcinoma: interim analysis of a cluster randomized controlled screening trial (PRO-NPC-001) in southern China. Ann Oncol. 2019 Oct 1;30(10):1630-1637. doi: 10.1093/annonc/mdz231. PMID 31373615
- [Background] Zhang MX, Li J, Shen GP, Zou X, Xu JJ, Jiang R, You R, Hua YJ, Sun Y, Ma J, Hong MH, Chen MY. Intensity-modulated radiotherapy prolongs the survival of patients with nasopharyngeal carcinoma compared with conventional two-dimensional radiotherapy: A 10-year experience with a large cohort and long follow-up. Eur J Cancer. 2015 Nov;51(17):2587-95. doi: 10.1016/j.ejca.2015.08.006. Epub 2015 Aug 26. PMID 26318726
- [Background] Zeng Y, Zhang LG, Wu YC, Huang YS, Huang NQ, Li JY, Wang YB, Jiang MK, Fang Z, Meng NN. Prospective studies on nasopharyngeal carcinoma in Epstein-Barr virus IgA/VCA antibody-positive persons in Wuzhou City, China. Int J Cancer. 1985 Nov 15;36(5):545-7. doi: 10.1002/ijc.2910360505. PMID 4055129
- [Background] Liu YP, Lv X, Zou X, Hua YJ, You R, Yang Q, Xia L, Guo SY, Hu W, Zhang MX, Chen SY, Lin M, Xie YL, Liu LZ, Sun R, Huang PY, Fan W, Guo X, Hong MH, Chen MY. Minimally invasive surgery alone compared with intensity-modulated radiotherapy for primary stage I nasopharyngeal carcinoma. Cancer Commun (Lond). 2019 Nov 15;39(1):75. doi: 10.1186/s40880-019-0415-3. PMID 31730020
- [Background] Chan KCA, Woo JKS, King A, Zee BCY, Lam WKJ, Chan SL, Chu SWI, Mak C, Tse IOL, Leung SYM, Chan G, Hui EP, Ma BBY, Chiu RWK, Leung SF, van Hasselt AC, Chan ATC, Lo YMD. Analysis of Plasma Epstein-Barr Virus DNA to Screen for Nasopharyngeal Cancer. N Engl J Med. 2017 Aug 10;377(6):513-522. doi: 10.1056/NEJMoa1701717. PMID 28792880
- [Background] Chan KC, Lo YM. Circulating EBV DNA as a tumor marker for nasopharyngeal carcinoma. Semin Cancer Biol. 2002 Dec;12(6):489-96. doi: 10.1016/s1044579x02000913. PMID 12450734